CLINICAL TRIAL: NCT03564938
Title: A Phase IV Study to Investigate the Safety and Efficacy of Regorafenib in Indian Patients With Metastatic Colorectal Cancer (mCRC).
Brief Title: Regorafenib in Indian Patients With Metastatic Colorectal Cancer (mCRC).
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19214
Record Dates: First submitted 2018-05-24; First posted 2018-06-21 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Colorectal Cancer
Keywords: mCRC
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regorafenib (Stivarga, BAY 73-4506) (Experimental): Patients with metastatic colorectal cancer
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — The recommended dose of regorafenib is 160 mg (consisting of 4 tablets, each containing 40 mg of regorafenib) for 3 weeks of every 4 week cycle, (ie. 3 weeks on therapy, 1 week off therapy).
  Other Names: Nublexa

SUMMARY:
This is a Phase IV, single-arm, prospective, open-label, multicenter, interventional study to evaluate safety and efficacy of regorafenib in patients with mCRC who have been previously treated with fluoropyrimidine , oxaliplatin-, and irinotecan based chemotherapy, an anti-VEGF therapy, and, if RAS wild type, an anti-EGFR therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients (≥18 years of age) with metastatic (Stage IV) colorectal adenocarcinoma confirmed either histologically or cytologically, with measurable metastatic disease according to RECIST v. 1.1
* Patients must have PD after receiving the approved standard therapies
* Patients must have ECOG PS of 0 or 1 and a life expectancy of at least 3 months
* Adequate bone marrow, liver and renal function
* Women of childbearing potential and men must agree to use adequate contraception

Exclusion Criteria:

* Unresolved toxicity greater than Grade 1 from prior treatment for mCRC
* Previous (within 28 days) or concomitant participation in another clinical study with investigational medicinal product(s)
* Subjects unable to swallow oral medications
* Any malabsorption condition
* Any medical or surgical conditions within 28 days before start of regorafenib that will interfere with patient's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | From the start of regorafenib treatment up to 30 days after the last dose of regorafenib
Changes in Eastern Cooperative Oncology Group Performance Status (ECOG PS) | From the start of regorafenib treatment up to 30 days after the last dose of regorafenib
Percentage of participants with change in worst grades for hematological and biochemical toxicities according to CTCAE version 4.03, based on laboratory measurements | From the start of regorafenib treatment up to 30 days after the last dose of regorafenib
Change in Body weight (kg) | From the start of regorafenib treatment up to 30 days after the last dose of regorafenib
Change in Body height (cm) | From the start of regorafenib treatment up to 30 days after the last dose of regorafenib
Change in Systolic / Diastolic BP (mmHg) | From the start of regorafenib treatment up to 30 days after the last dose of regorafenib
Change in heart rate (beats/min) | From the start of regorafenib treatment up to 30 days after the last dose of regorafenib

SECONDARY OUTCOMES:
Disease control rate (DCR) | In each participant, every 8 weeks from the start of regorafenib until radiological disease progression, lost to follow-up, consent withdrawn or end of study, whichever occurs first
  Defined as proportion of patients achieving complete response (CR), partial response (PR), or SD (stable disease) per Response Evaluation Criteria in Solid Tumors (RECIST) v. 1.1
Overall response rate (ORR) | In each participant, every 8 weeks from the start of regorafenib until radiological disease progression, lost to follow-up, consent withdrawn or end of study, whichever occurs first
  Defined as proportion of patients achieving CR, and PR per RECIST v.1.1
Progression free survival (PFS) | In each participant, every 8 weeks from the start of regorafenib until radiological disease progression, lost to follow-up, consent withdrawn or end of study, whichever occurs first
  Progression free survival is defined as the time from study drug assignment to progressive disease (PD) or death from any cause or date of last tumor assessment if the patient did not progress or die.
Overall survival (OS) | In each participant, every 8 weeks from the start of regorafenib until death, lost to follow-up, consent withdrawn or end of study, whichever occurs first
  Overall survival is defined as the time from study drug assignment to death from any cause or last date when the patient was known to be alive.

CONTACTS AND LOCATIONS:
Locations (13):
- India (13):
  - Apollo Research Foundation, Hyderabad, Andhra Pradesh
  - Shalby Hospital, Ahmedabad, Gujarat
  - Healthcare Center Global Hospital, Ahmedabad, Gujarat
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - Jaslok Hospital and Research Centre, Mumbai, Maharashtra
  - Sushrut Hospital & Research Centre, Mumbai, Maharashtra
  - Jehangir Hospital, Pune, Maharashtra
  - Fortis Hospital, West-Mumbai, Maharashtra
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Sparsh Hospital & Critical Care, Bhubaneswar, Odisha
  - Apollo Speciality Hospitals, Madurai, Tamil Nadu
  - IPGME & R / SSKM Hospital, Kolkata, West Bengal
  - Health Point Hospital, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, they study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/19214
- See also: Study_Synopsis-19214.docx attachment has been generated from the Study Synopsis template. Data may be populated from the following (as available) : Study (255.0), Protocol (38.2), Results(0.1) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217261&parentIdentifier=19214&attachmentIdentifier=0bcd1efc-e45e-4f5d-bc72-fd89716bf3af&fileName=19214_Websynopsis_CTP.pdf&versionIdentifier=